CLINICAL TRIAL: NCT02726425
Title: Women in Control: A Virtual World Study of Diabetes Self-Management. Translational Research to Improve Diabetes and Obesity Outcomes (R01)
Brief Title: Women in Control: A Virtual World Study of Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: University of Massachusetts, Worcester (Other); Boston University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-34220; 1R01DK106531 (NIH)
Record Dates: First submitted 2016-03-28; First posted 2016-04-01 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes self management; Second Life platform; Medical group visits
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Life Participants (Experimental): Half of participants will receive the Diabetes Self Management Medical Group Visits intervention while meeting in the virtual world (Second Life platform)
  Interventions: Behavioral: Diabetes Self Management Medical Group Visits
- Face-to-Face Participants (Active Comparator): The other half of the participants will receive the Diabetes Self Management Medical Group Visitsintervention while meeting face-to-face in person at Boston Medical Center.
  Interventions: Behavioral: Diabetes Self Management Medical Group Visits

INTERVENTIONS:
Behavioral: Diabetes Self Management Medical Group Visits — The Women in Control DSM intervention involves: (1) 8-wk series of interactive, educational medical group visit sessions with groups of 10-12 participants, led by clinicians & peer leaders lasting ~100'' in length conducted either in Spanish or English and (2) Individual consultation with a clinician lasting 10-15 minutes. Group visits will consist of experiential and discussion based learning of topics including the importance of diet, physical activity, medications, mindfulness and stress reduction to diabetes self management.

SUMMARY:
This study evaluates the comparative effectiveness of a diabetes self management (DSM) group medical visit in the virtual world (Second life) verses a face-to-face format, aimed to increase physical activity and improve glucose control among Black/African American and Hispanic women with uncontrolled diabetes mellitus.

DETAILED DESCRIPTION:
The prevalence of diabetes mellitus (DM) in the US is disproportionately high among minority women. In order to participate as partners in healthcare, DM patients need self-management education and support. Diabetes self-management (DSM) support is effective in helping DM patients make good choices and achieve clinical goals but is difficult to deliver in medical practice settings. Virtual reality technology can assist DM patients and their clinical teams with DSM support by providing effective educational tools in an engaging, learner-centered context that fosters self-efficacy and skill proficiency. Our prior work demonstrated that virtual worlds, like Second Life (SL), are suitable for supporting DSM education for patients. SL, an Internet-based virtual world, is an example of an immersive, three-dimensional environment which supports social networking and interaction with information.

The investigators now aim to enhance the existing diabetes curriculum using a medical group visit design to study whether the Women in Control virtual world group medical visit leads to similarly effective health and educational outcomes compared to face-to-face group medical visits. The investigators aims are to conduct a randomized, controlled trial of the comparative effectiveness of a virtual world DSM group medical visit format vs. a face-to-face DSM group visit format to increase physical activity and improve glucose control among Black/African American and Hispanic women with uncontrolled DM at six month follow up, and to conduct a qualitative, ethnographic study of participant engagement with the virtual world platform during the virtual world group sessions, between group sessions, and following completion of the eight-week curriculum to characterize learners' self-directed interactions with the technology platform and assess the correlation of these interactions with DSM behaviors and diabetes control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus (documented in the medical chart)
* Last recorded HbA1c >8.0
* Currently treated with diet, oral hypoglycemic agents or insulin
* Black/African American or Hispanic/Latina origin
* Has telephone access
* Able to understand and participate in study protocol
* Functionally capable of meeting the activity goals
* Understand and give informed consent
* Physician approval to participate in study
* Can communicate in English or Spanish

Exclusion Criteria:

* History of diabetic ketoacidosis
* Currently or planning pregnancy
* Unable or unwilling to provide informed consent
* Plans to leave area within 6 month study period that would interfere with ability to attend 8 weekly sessions and/or 6 month follow up
* Required intermittent glucocorticoid therapy within past 3 months.
* Experienced acute coronary event (myocardial infarction or unsable angina) within previous 6 months
* Medical condition that precludes adherence to study dietary recommendations (i.e. Crohn's, ulcerative colitis, etc)
* Medical or serious psychiatric illness (dementia, suicidal within last 5 months, psychiatric hospitalization). Those with diagnosis of depression or who take antidepressents are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2015-07; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in physical activity level | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Participants will wear an activity monitor for a week at each collection point. Results measured in METs/hr.
Change in disease control (HbA1c) | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Change in HbA1c from BMC laboratory blood testing results

SECONDARY OUTCOMES:
Patient Activation | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Measured by change in PAM 13 score
Medication Adherence | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Prescription fulfillment ratio per i2b2 database claims data analysis
Depression | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Change in Patient Health Questionnaire (PHQ8) score
Improvement in cholesterol, hypertension and body weight | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Serum LDL/HDL from BMC laboratory results. BP from home blood pressure monitor readings. BMI from weight/height measurements.
Health-Related Quality of Life | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Change in Q-LES-Q screening survey
Dietary Habits | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Multiple measures of 24-hr dietary recall
Functional Status | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Measured by Sheehan disability scale
Stress | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Measured by perceived stress scale (PSS-10)
Social Support | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Measured by MOS social support survey
Health Service Utilization | Data collection at baseline, post-intervention (8 weeks) and at 6 months follow up
  Self-report and chart review of hospitalizations, PCP and specialist visits

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E Mitchell, MD, MS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell SE, Mako M, Sadikova E, Barnes L, Stone A, Rosal MC, Wiecha J. The comparative experiences of women in control: diabetes self-management education in a virtual world. J Diabetes Sci Technol. 2014 Nov;8(6):1185-92. doi: 10.1177/1932296814549829. Epub 2014 Sep 10. PMID 25212580
- [Derived] Mitchell SE, Bragg A, De La Cruz BA, Winter MR, Reichert MJ, Laird LD, Moldovan IA, Parker KN, Martin-Howard J, Gardiner P. Effectiveness of an Immersive Telemedicine Platform for Delivering Diabetes Medical Group Visits for African American, Black and Hispanic, or Latina Women With Uncontrolled Diabetes: The Women in Control 2.0 Noninferiority Randomized Clinical Trial. J Med Internet Res. 2023 May 10;25:e43669. doi: 10.2196/43669. PMID 37163341